CLINICAL TRIAL: NCT06636591
Title: A Prospective, Open-label, Single-center, Pilot Study of Neoadjuvant Chemotherapy Combined With Immunotherapy and Multimodal Thermal Therapy for HER2-negative Breast Cancer
Brief Title: Pilot Study of Neoadjuvant Chemotherapy Combined With Immunotherapy and Multimodal Thermal Therapy for HER2-negative Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MTT-BC-002
Record Dates: First submitted 2024-09-29; First posted 2024-10-10 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer Female; HER2-negative Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Triple-negative Breast Cancer with Non-immunomodulatory Subtype (Experimental)
  Interventions: Combination Product: Device: Multimodal Tumor Thermal Therapy System Drug: Camrelizumab Drug: Nab paclitaxel Drug: Carboplatin
- Hormone Receptor-positive (HR+) and HER2-negative (HER2-) (Experimental)
  Interventions: Combination Product: Device: Multimodal Tumor Thermal Therapy System Drug: Camrelizumab Drug: Nab paclitaxel Drug: Carboplatin Drug: Goserelin

INTERVENTIONS:
Combination Product: Device: Multimodal Tumor Thermal Therapy System Drug: Camrelizumab Drug: Nab paclitaxel Drug: Carboplatin — Drugs was given a few days after multimodal thermal therapy
  Arms: Triple-negative Breast Cancer with Non-immunomodulatory Subtype
Combination Product: Device: Multimodal Tumor Thermal Therapy System Drug: Camrelizumab Drug: Nab paclitaxel Drug: Carboplatin Drug: Goserelin — Drugs was given a few days after multimodal thermal therapy
  Arms: Hormone Receptor-positive (HR+) and HER2-negative (HER2-)

SUMMARY:
In this study, breast cancer (BC) patients eligible for inclusion will be divided into two groups according to molecular typing and subtyping, which combined immunotherapy and multimodal thermal therapy with conventional neoadjuvant chemotherapy, to explore methods of immune induction for BC, enhance the efficacy of immunotherapy, and accumulate data for subsequent stages of clinical study.

DETAILED DESCRIPTION:
Local tumor destruction with non-surgical ablation (NSA, cryoablation or radiofrequency) induces inflammation and releases antigens that can activate tumor-specific immune responses.

Pre-clinically, we demonstrated that multimodal thermal therapy (MTT) as an integrated treatment modality of cryotherapy and radiofrequency heating, can effectively activate systemic and long-lasting antitumor immunity.

In this pilot study, patients with operable HER2-negative breast cancer were designed to receive a combination of MTT, immunotherapy and neoadjuvant chemotherapy. Potential favorable intra-tumoral and systemic immunologic effects were assessed with the combination, revealing the possibility for induced and synergistic anti-tumor immunity with this strategy.

ELIGIBILITY:
Inclusion Criteria:

1. Female，age 18-70 years.
2. Histologically confirmed invasive cancer of the breast, and patients meeting cT2-4N+M0 criteria;
3. TNBC non-immunoregulation subtype or HR+/HER2- status were measured by immunohistochemistry (IHC);
4. At least one measurable lesion according to RECIST 1.1 criteria;
5. Normal organ and marrow function: Hemoglobin (HB) ≥90 g/L (No blood was transfused within 14 days), Absolute neutrophil count ≥ 1500/μL, Platelets ≥ 75,000/μL, Total bilirubin ≤ 1.5 x ULN), aspartate aminotransferase (AST) (SGOT) and alanine aminotransferase (ALT) (SGPT) ≤ 3 x ULN, creatinine < 1 x ULN, endogenous creatinine clearance > 50 ml/min (Cockcroft-Gault formula);
6. LVEF ≥55%;
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
8. Non-pregnant and non-lactating, fertile female subjects were required to use a medically approved contraceptive method for the duration of the study treatment and at least 3 months after the last use of the study drug;
9. Ability to understand and willingness to sign a written informed consent.

Exclusion Criteria:

1. Previous cytotoxic chemotherapy, endocrine therapy, biological therapy or radiotherapy for any reason;
2. Patients with New York Heart Association (NYHA) grade II or above heart disease (including grade II);
3. Patients with severe systemic infections or other serious diseases;
4. Patients with known allergy or intolerance to the study drug or its excipients;
5. Other malignant tumors in the past 5 years, except cured cervical carcinoma in situ and non-melanoma skin cancer;
6. Pregnant or lactating patients of childbearing age who refused to take appropriate contraceptive measures during the course of the study;
7. Participated in other trial studies within 30 days before the administration of the first dose of the study drug;
8. Endocrine system disorders;
9. Patients who were judged by the investigator to be unsuitable for this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2024-11-18 (Estimated); Primary Completion 2025-02-07 (Estimated); Study Completion 2026-10-07 (Estimated)

PRIMARY OUTCOMES:
Assessment of immune activating response | up to 28 weeks
  * Proportion of subjects with immune response to combination therapy detected by biomarkers in peripheral blood samples
  * Evaluate the infiltration of immune cells in tumor areas and adjacent tissues

SECONDARY OUTCOMES:
CTCAE scale (V4.0) | up to 28 weeks
  To evaluate the rate of adverse effects of patient by the standard CTCAE scale (V4.0)

CONTACTS AND LOCATIONS:
Locations (1):
- Breast cancer institute of Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China